CLINICAL TRIAL: NCT04560088
Title: Mindfulness Training to Reduce Social Isolation and Feelings of Loneliness in Older Caregivers for Family Members With Alzheimer's Disease and Related Dementias
Brief Title: Mindfulness to Reduce Loneliness in Older Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Autumn Gallegos, Assistant Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5296; P30AG064103 (NIH)
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Social Isolation; Loneliness
Keywords: Mindfulness; Caregiver; Alzheimer's Disease; Dementia
MeSH Terms: conditions — Social Isolation; Alzheimer Disease; Dementia | interventions — Mindfulness; Respiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Mindfulness using an individual mobile health mindfulness-based intervention training. These sessions are intended to act as a general introduction to mindfulness meditation and incorporate techniques such as breath awareness and body scanning.
  Interventions: Behavioral: Mindfulness
- Breathing (Active Comparator): Breathing control intervention will use an individual breathing app. The intervention is designed to be structurally equivalent to the mindfulness-based study intervention on key common factors of psychosocial interventions: (a) the number of sessions, (b) the length of sessions, and (c) delivery format.
  Interventions: Behavioral: Breathing

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness-based mobile health intervention.
  Arms: Mindfulness
Behavioral: Breathing — Breathing mobile health intervention.
  Arms: Breathing

SUMMARY:
The objective of this pilot study is to provide initial evidence of the role of mindfulness training in improving social disconnectedness - including social isolation and feelings of loneliness - in older caregivers for family members with ADRD. The investigators propose a two-arm randomized control trial: participants will be randomized to (a) smartphone-based MBSR app (Headspace) or (b) active control (breathing app) for 14 days. Loneliness and quality of social interactions will be assessed using Ecological Momentary Assessment at baseline and 14-days after randomization.

DETAILED DESCRIPTION:
Social isolation and feelings of loneliness are risk factors for older caregivers for family members with Alzheimer's Disease and Related Dementias (ADRD). Further, social isolation and loneliness place older caregivers at risk of poor health, including increased inflammation, cardiovascular disease, depression, and premature mortality. Interventions to promote social connectedness in older caregivers have the potential to reduce elevated morbidity and premature mortality and buffer the high caregiving burden in this growing but understudied population. Thus, developing effective treatments to reduce social disconnectedness in older adults is essential, but previous behavioral treatment efforts have had limited success. Mindfulness-based interventions may reduce loneliness in older adults, as demonstrated in a randomized controlled trial of an 8-week mindfulness-based stress reduction program. Another recent study demonstrated the efficacy of a smartphone-based mindfulness training for reducing loneliness and increasing social contact in daily life among adults reporting above average stress; however, smartphone-based mindfulness training interventions have not been tested with older adults, nor have they been tested with caregivers of family members with ADRD. Specifically, prior studies were conducted with healthy adults not necessarily burdened by caregiving; it remains unknown how caregiver stress --related to competing demands on time and significant loneliness --may impact the ability to comply with the intervention as well as indicate barriers to efficacy. The current study will follow a similar protocol as the aforementioned randomized controlled trial that used a smartphone-based mindfulness training to address loneliness and social contact.

ELIGIBILITY:
Inclusion Criteria:

* English speaking.
* Caregiver for a community-dwelling family member with ADRD, living with (or in close proximity to) family member with dementia.
* Elevated caregiving distress: above population mean (>11) on 10-item Perceived Stress Scale (PSS-10) and/or at least moderate caregiver strain (score >= 5) on the Modified Caregiver Strain Index (MCSI).
* Social disconnectedness: UCLA Loneliness Scale: Short Form score of >6 (except for n=5 in Aim 1 who report feeling socially connected).
* Access to e-mail in order to complete the e-consent module in REDCap which will be used in this study.

Exclusion Criteria:

* Non-English speaking because our primary community partner agency (Lifespan) cannot currently accommodate non-English speaking clients.
* Current problem drinking will be assessed using the AUDIT-C during the phone screen (score of 5 or greater indicating exclusion).
* Modules from the Mini International Neuropsychiatric Exam (MINI) will be used to exclude subjects who have these psychiatric conditions: current non-alcohol psychoactive substance abuse, psychotic disorders (current and lifetime), bipolar disorder, and current mood disorder with psychotic features.
* Those with significant cognitive impairment on a cognitive screening measure at the HARP screening assessment.
* In order to test the effects of developing mindfulness skills in a novice population, those with a regular systematic mindfulness meditation or related mind-body practice (>2 times per week) will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Autumn Gallegos, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Gallegos AM, Chapman BP, Kaplan J, Van Orden KA, Heffner KL. A pilot randomized mobile health mindfulness intervention for older adult caregivers of family members with Alzheimer's disease and related dementias. Aging Ment Health. 2025 Dec;29(12):2165-2172. doi: 10.1080/13607863.2025.2506774. Epub 2025 May 28. PMID 40435371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness | Breathing
Started | 24 | 31
Completed | 19 | 30
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Breathing | Total
Number analyzed (Participants) | 24 | 31 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 19 | 33
  >=65 years | 10 | 12 | 22
Age, Continuous [Mean (Full Range); unit: years] | 65 [52 to 81] | 64 [51 to 85] | 64 [51 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 31 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 22 | 28 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 31 | 55

OUTCOME MEASURES:

1. Primary Outcome: Five Facet Mindfulness Questionnaire (FFMQ)
Description: The FFMQ assesses five factors that represent mindfulness as it is currently conceptualized: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience, and a total score indicating overall mindfulness. The 39 items of the FFMQ are rated on a 5-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true). The total score ranges from 39-195, with higher scores indicating greater mindfulness. Data presented is for the total FFMQ score.
Time Frame: 20 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness | Breathing
Number analyzed (Participants) | 24 | 31
score on a scale
  Baseline (Time 1) | 137.83 (21.92) | 127.81 (20.01)
  Day 20 (Time 2) | 137.42 (20.19) | 134.32 (21.99)

2. Primary Outcome: Difficulties in Emotion Regulation Scale (DERS)
Description: The DERS is a 36-item self-report measure that assesses emotion dysregulation in six domains: nonacceptance of emotional responses, difficulties engaging in goal directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. The DERS has demonstrated high internal consistency in clinical and nonclinical samples, good test-retest reliability over 8-weeks, construct validity, and sensitivity to change over time following interventions, including acceptance and mindfulness therapies. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Scores range from 36-180, with higher scores indicating more difficulty in emotion regulation. Data presented is for the total DERS score.
Time Frame: 20 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness | Breathing
Number analyzed (Participants) | 24 | 31
score on a scale
  Baseline (Time 1) | 67.25 (17.68) | 86.45 (25.11)
  Day 20 (Time 2) | 70.32 (26.85) | 78.19 (22.67)

3. Primary Outcome: The UCLA 3-Item Loneliness Scale
Description: This assessment has demonstrated excellent internal consistency, test re-test reliability, and construct validity (associations with social support, social network size). Each question is rated on a 3-point scale: 1 = Hardly Ever; 2 = Some of the Time; 3 = Often. All items are summed to give a total score, ranging from 3-9 points. Higher scores indicate more loneliness.
Time Frame: 20 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness | Breathing
Number analyzed (Participants) | 24 | 31
score on a scale
  Baseline (Time 1) | 6.04 (1.92) | 7 (1.73)
  Day 20 (Time 2) | 6.44 (1.92) | 6.35 (1.70)

ADVERSE EVENTS:
Time Frame: 20 days
Arm/Group | Mindfulness | Breathing
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/31
Other Adverse Events (participants affected / at risk) | 0/24 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness (N=24) | Breathing (N=31)
Interpersonal threat (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT04560088/Prot_SAP_000.pdf